CLINICAL TRIAL: NCT03245411
Title: A Randomized, Controlled Trial to Assess Multi-Level Interventions to Improve Adherence to Oral Medications in Cancer Patients in a Socioeconomically Disadvantaged Community
Brief Title: Assessment of Multi-Level Interventions to Improve Adherence to Oral Medications in Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 4950; JT 27684 (Other: JeffTrial Number)
Record Dates: First submitted 2017-08-02; First posted 2017-08-10 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial (RCT) Single Center
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care (Control Group) (No Intervention): All participants in this group will receive the standard of care intervention provided by the RN.
- Intervention Group (Experimental): In addition to the standard of care, the participants randomized to Intervention Group will be invited to a separate room. The following activities will be undertaken, in order to address patients' questions and concerns, and discuss potential solutions to their barriers to care
  The patient will be asked to watch brief educational videos on "Life with oral cancer treatment." The information contained in the videos will be reinforced with materials written at a 4th grade level, that correspond to each of the brief videos.The patient will receive a brief phone call (from the study coordinator) on the first business day following the baseline interview, and thereafter, two weeks following each visit to the oncology clinic.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — All participants in this group will receive the standard of care intervention provided by the RN. This includes:Education in the clinic setting,Printed information about the chemotherapy drug and chemotherapy side effects. The RN will be blinded to the arm of study to which each patient is allocated.
  Arms: Intervention Group

SUMMARY:
Einstein Medical Center in Philadelphia serves a diverse group of the patient population. The majority of patients have a diverse cultural background, low literacy, and poor social-economic status. Medication adherence for chronic medical problems is in a range of 40-70%. Medication adherence among patients on oral anti-cancer therapy is not studied in detail. The main objective is to study medication adherence to oral anticancer agents in patients with low literacy and poor socio-economic status.

DETAILED DESCRIPTION:
Until recently, contemporary approaches to cancer care have failed to consistently tailor communication approaches to patients with low health literacy. They have produced mixed results in regard to implementation of successful interventions in addressing the needs of this populations. Low health literacy is especially common in medically underserved communities, including in North Philadelphia. Cancer treatment, including cancer chemotherapy, is complex, and it requires substantial skills, in order for patients to adhere to care and achieve the goals of therapy. Patients with low health literacy find it especially challenging to navigate cancer treatment. Results of previous research showed that intervention strategies that address the needs for information and material support of African American older adults, can help improve adherence to cancer screening in this population.

The purpose is to develop and evaluate model interventions to improve healthcare outcomes for socially disadvantaged populations. The objective in this proposal is to conduct a randomized controlled trial that evaluates the effects of an intervention that provides enhanced education and material support, on adherence to care, among the cancer patients of the Medical Oncology Clinic of the Einstein Medical Center in Philadelphia.

The central hypothesis is that compared to the standard educational intervention delivered by a registered nurse, the addition of an enhanced intervention (enhanced education, problem-solving skills and facilitative support) will result in greater adherence care, especially among patients with low health literacy.

ELIGIBILITY:
Inclusion Criteria:

* All patients on oral chemotherapeutic agents
* Clinical diagnosis of stage IV breast cancer
* Clinical diagnosis of stage III and IV colorectal cancer (not receiving concurrent radiation therapy)
* Clinical diagnosis of stage IV non-small cell lung cancer
* Clinical diagnosis of stage IV renal cell carcinoma
* Clinical diagnosis of stage IV ovarian carcinoma
* Clinical diagnosis of multiple myeloma
* Clinical diagnosis of chronic myelogenous leukemia on TKI
* Clinical diagnosis of myelodysplastic syndrome on Lenalidomide
* Adjuvant treatment for Gastro Intestinal Stromal Tumor
* Clinical diagnosis of chronic Lymphocytic Leukemia
* Clinical diagnosis of metastatic Prostate cancer
* Clinical diagnosis of hepatocellular Carcinoma
* Clinical diagnosis of stage IV Melanoma
* Clinical diagnosis of myelofibrosis/myeloproliferative neoplasms
* Age >18 years
* ECOG Performance Status <3

Exclusion Criteria:

* ECOG Performance Status of 3 and above
* Concurrent chemo radiation
* Non-English speaker
* Clinical diagnosis of dementia, or otherwise unable to give informed consent.
* History of non-compliance (defined as the history of 2 or more missed appointments in the clinic).
* Pregnant patients
* Nursing Home Patients
* Incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2025-12-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Adherence to oral chemotherapy | 6 months
  Frequency of missed chemotherapy doses post randomization (based on interviews)

SECONDARY OUTCOMES:
Frequency of medication refills | 6 months
  Prescription refills, based on pharmacy records
Adherence to scheduled follow-up medical care visits | 6 months
  Frequency and adherence to schedule follow up visit
Healthcare utilization | 6 months
  Any unscheduled visit (office Visit, ED Visits, Hospitalization, use of preventive care)

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Dourado, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Albert Einstein Healthcare Network, Philadelphia, Pennsylvania, United States